CLINICAL TRIAL: NCT02311894
Title: A Phase IV, Multicenter, Open-Label Study of the Immunogenicity of Nutropin AQ® V1.1 [Somatropin (rDNA Origin) Injection] Administered Daily to Naïve Growth Hormone-Deficient Children (iSTUDY)
Brief Title: A Post-Marketing Study of the Immunogenicity of Somatropin (Ribosomal Deoxyribo Nucleic Acid [rDNA] Origin) Injection (Nutropin AQ®) in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29543
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental): Children will receive daily SC injections of somatropin at a dose of up to 0.043 milligrams per kilogram per day (mg/kg/day) for 1 year.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Somatropin will be administered as SC injections at a dose of up to 0.043 mg/kg/day. The dose may be adjusted for a change in body weight of at least (plus [+]/minus [-]) 2 kilograms (kg) from baseline at the Month 6 study visit or for a change in insulin-growth factor-1 (IGF-1), as per investigator assessment.
  Other Names: Nutropin AQ v1.1

SUMMARY:
This is a Phase IV, multicenter, open-label, single-arm study of somatropin (rDNA origin) (Nutropin AQ v1.1) in pre-pubertal children with growth hormone deficiency (GHD) naïve to prior recombinant human growth hormone (rhGH) treatment. The study is designed to characterize the immunogenicity profile of somatropin (rDNA origin) injection when administered daily subcutaneously for 12 months. The clinical impact of immunogenicity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Bone age less than equal to (</=) 9 years (females) or </= 11 years (males) as determined by X-ray of the left hand and wrist using Greulich and Pyle method and obtained within the 12 months prior to enrollment
* Prepubertal (Tanner I) males and females by physical examination
* Diagnosis of GHD (stimulated GH less than [<] 10 nanograms per milliliter [ng/mL]) by two standard pharmacologic tests obtained up to 12 months prior to informed consent/assent
* Normal thyroid function test within the 12 months prior to informed consent/assent
* Normal complete blood counts within 12 months prior to informed consent/assent
* Documentation of prior height and weight measurements, with height standard deviation score (SDS) </= 5th percentile for idiopathic isolated GHD participants

Exclusion Criteria:

* Any previous rhGH treatment
* Short stature etiologies other than GHD
* Acute critical illness or uncontrolled chronic illness, which in the opinion of the investigator and medical monitor, would interfere with participation in this study, interpretation of the data, or pose a risk to participant safety
* Chronic illnesses such as inflammatory bowel disease, celiac disease, heart disease, and diabetes
* Bone diseases such as achondroplasia or hypochondroplasia, intracranial tumor, irradiation, and traumatic brain injury
* Participants receiving oral or inhaled chronic corticosteroid therapy (greater than [>] 3 months) for other medical conditions other than central adrenal insufficiency
* Participants who require higher (2 times or greater than maintenance) doses of corticosteroids for more than 5 days in the 6 months prior to enrollment in the study
* Participants with active malignancy or any other condition that the investigator believes would pose a significant hazard to the participant if rhGH were initiated
* Females with Turner syndrome regardless of their GH status
* Prader-Willi syndrome regardless of GH status
* Born small for gestational age regardless of GH status
* Presence of scoliosis requiring monitoring
* Previous participation in another clinical trial or investigation of GH, treatment for growth failure, or treatment with a biologic agent
* Participants with closed epiphyses
* Participants with a known hypersensitivity to somatropin, excipients, or diluent

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (33):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Children'S Hospital of Orange County, Orange, California
  - Center of Excellence in Diabetes & Endocrinology, Sacramento, California
  - San Diego Medical Group; Pediatric Endocrinology, San Diego, California
  - Rocky Mountain Pediatric Endocrinology, PC, Centennial, Colorado
  - Pediatric Endocrine Associates, Greenwood Village, Colorado
  - Nemours Children's Clinic - of the Nemours Foundation, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Nemours Childrens Clinic, Orlando, Florida
  - The Pediatric Endocrine Office of Larry C. Deeb, Tallahassee, Florida
  - Pediatric Endrocine Assoc, Tampa, Florida
  - USF Diabetes Center, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Barry J Reiner, MD, LLC, Baltimore, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - Baystate Endocrinology and Diabetes; Baystate Children's Specialty Center, Pediatric Endocrinology, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Childrens' Hospital, Minneapolis, Minnesota
  - Children's Healthcare d.b.a Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - Children's Mercy Hospitals & Clinics; Pulmonology, Kansas City, Missouri
  - Hackensack University Medical Center PARTNER, Hackensack, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - UNC General Pediatrics Clinic, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Milton S Hershey Ped Sub Spclt, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina; MUSC Pediatric Endocrinology, Charleston, South Carolina
  - Endocrine Associates of Dallas, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin: Children will receive daily subcutaneous (SC) injections of somatropin at a dose of up to 0.043 milligrams per kilogram per day (mg/kg/day) for 1 year.
Period: Overall Study
Arm/Group | Somatropin
Started | 82
Modified ITT Population (Participants who took at least one dose of study drug and had at least one post-baseline assessment.) | 81
Completed | 78
Not Completed | 4
Not completed — Discontinued in error | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Somatropin
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5
  Black or African American | 2
  Multiple | 1
  Other | 3
  Unknown | 3
  White | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Develop Anti-GH Antibodies After Treatment With Nutropin AQ v1.1
Description: Participants who were tested positive to anti-GH antibody after initiation of study treatment.
Time Frame: Baseline up to 1 year
Population: All enrolled participants who received at least one dose of study drug and who had at least one post-baseline assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Somatropin
Number analyzed (Participants) | 81
percentage of participants | 3.7 [0.77 to 10.44]

2. Secondary Outcome: Percentage of Participants Who Exhibit Functional Growth Attenuation
Description: Growth attenuation is defined as initial growth response greater than pretreatment velocity followed by reduction in growth response to below the pretreatment velocity in the subsequent 6- to 12-month treatment period or reaching ≤ 2 cm per year.
Time Frame: Baseline up to 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Somatropin
Number analyzed (Participants) | 81
percentage of participants | 2.6 [0.31 to 8.96]

3. Secondary Outcome: Percentage of Participants With Neutralizing Antibodies
Description: Among participants who developed positive anti-GH antibody post-baseline, participants who were tested positive to neutralizing anti-GH antibody during study participation.
Time Frame: Baseline up to 1 year
Population: Included only patients who had positive anti-GH antibody.
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin
Number analyzed (Participants) | 3
percentage of participants | 0

4. Secondary Outcome: Annualized Growth Velocity at Months 6 and 12 (Change From Baseline)
Description: Annualized growth velocity is defined as (height - baseline height) / (date of height assessment - date of baseline)*365.25. Results are presented according to anti-GH antibody status (positive included all participants that were anti-GH antibody positive at least once post-baseline visit and anti-GH antibody negative population included all participants that were anti-GH antibody negative at all post-baseline visits).
Time Frame: Months 6, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Somatropin
Number analyzed (Participants) | 81
cm/year
  6 months (Anti-GH Antibody Positive): number analyzed (Participants) | 3
  6 months (Anti-GH Antibody Positive) | 5.3 (2.89)
  6 months (Anti-GH Antibody Negative): number analyzed (Participants) | 67
  6 months (Anti-GH Antibody Negative) | 5.5 (2.64)
  12 months (Anti-GH Antibody Positive): number analyzed (Participants) | 2
  12 months (Anti-GH Antibody Positive) | 5.2 (3.61)
  12 months (Anti-GH Antibody Negative): number analyzed (Participants) | 57
  12 months (Anti-GH Antibody Negative) | 4.9 (2.40)

5. Secondary Outcome: Height Standard Deviation Score (SDS) at Months 6 and 12 (Change From Baseline)
Description: Height Standard Deviation Score (SDS) allows for the comparison of a participants height to that of others in the same age group. Therefore, the average height for that age group will have the SDS of 0. In this study, the starting Height SDS score was ≤ -1.5 (≤ 5th percentile). Results are presented according to anti-GH antibody status (positive included all participants that were anti-GH antibody positive at least once post-baseline visit and anti-GH antibody negative population included all participants that were anti-GH antibody negative at all post-baseline visits.
Time Frame: Months 6, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Somatropin
Number analyzed (Participants) | 81
SDS
  6 months (Anti-GH Antibody Positive): number analyzed (Participants) | 3
  6 months (Anti-GH Antibody Positive) | 0.3 (0.11)
  6 months (Anti-GH Antibody Negative): number analyzed (Participants) | 67
  6 months (Anti-GH Antibody Negative) | 0.4 (0.17)
  12 months (Anti-GH Antibody Positive): number analyzed (Participants) | 2
  12 months (Anti-GH Antibody Positive) | 0.8 (0.15)
  12 months (Anti-GH Antibody Negative): number analyzed (Participants) | 57
  12 months (Anti-GH Antibody Negative) | 0.7 (0.25)

6. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Among participants who received at least one dose of study drug, those who reported at least one adverse event during study participation.
Time Frame: Baseline up to 1 year
Population: Include all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Somatropin
Number analyzed (Participants) | 82
percentage of participants | 69.5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from Day 1 until 28 days after last dose of study medication for up to 12 months.
Description: The safety population included all participants who received at least 1 dose of the investigational product.
Arm/Group | Somatropin
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 40/82
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin (N=82)
Vomiting (Gastrointestinal disorders) | 12
Injection site bruising (General disorders) | 7
Pyrexia (General disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 8
Pharyngitis streptococcal (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 5
Headache (Nervous system disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT02311894/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02311894/SAP_001.pdf